CLINICAL TRIAL: NCT04139798
Title: A Phase 3, Multi-Center, Randomized, Double-Masked, Saline-Controlled Trial to Evaluate the Effect of NOV03 (Perfluorohexyloctane) on Signs and Symptoms of Dry Eye Disease Associated With Meibomian Gland Dysfunction (Gobi Study)
Brief Title: Perfluorohexylcotane (NOV03) for the Treatment of Signs and Symptoms of Dry Eye Disease Associated With Meibomian Gland Dysfunction (Gobi Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NVU-003 (Gobi)
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NOV03 4 times daily (QID) (Experimental): 100% Perfluorohexyloctance solution 4 times daily (QID)
  Interventions: Drug: NOV03
- Placebo 4 times daily (QID) (Placebo Comparator): Saline solution (0.6% sodium chloride solution) 4 times daily (QID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NOV03 — 100% Perfluorohexyloctane
  Arms: NOV03 4 times daily (QID)
Drug: Placebo — Saline solution (0.6% sodium chloride solution)
  Arms: Placebo 4 times daily (QID)

SUMMARY:
This trial will evaluate the efficacy, safety, and tolerability of NOV03 ophthalmic solution in comparison to a saline control for the treatment of the signs and symptoms of Dry Eye Disease (DED) associated with Meibomian Gland Dysfunction (MGD).

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF (Informed Consent Form)
* Subject-reported history of Drye Eye Disease (DED) in both eyes
* Ability and willingness to follow instructions, including participation in all study assessments and visits

Exclusion Criteria:

* Women who are pregnant, nursing or planning pregnancy
* Unwillingness to submit a blood pregnancy test at screening and the last visit (or early termination visit) if of childbearing potential, or unwillingness to use acceptable means of birth control
* Clinically significant slit-lamp findings or abnormal lid anatomy at screening and Visit 1
* Ocular/peri-ocular malignancy
* History of herpetic keratitis
* Active ocular allergies or ocular allergies that are expected to be active during the study
* Ongoing ocular or systemic infection
* Wear contact lenses within 1 month prior to screening or anticipated use of contact lenses during the study
* Intra-ocular surgery or ocular laser surgery within the previous 6 months, or have planned ocular and/or lid surgeries over the study period
* Presence of uncontrolled systemic diseases
* Presence of known allergy and/or sensitivity to the study drug or saline components
* Use of any topical steroids treatments, topical cyclosporine, lifitegrast, serum tears or topical anti-glaucoma medication within 2 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Bausch Health
Locations (29):
- United States (29):
  - Bausch Site 124, Birmingham, Alabama
  - Bausch Site 125, Scottsdale, Arizona
  - Bausch Site 110, Glendale, California
  - Bausch Site 121, Long Beach, California
  - Bausch Site 102, Mission Hills, California
  - Bausch Site 101, Newport Beach, California
  - Bausch Site 116, Rancho Cordova, California
  - 103, Torrance, California
  - Bausch Site 123, Torrance, California
  - Bausch Site 127, Danbury, Connecticut
  - Bausch Site 129, Fort Myers, Florida
  - Bausch Site 115, Jacksonville, Florida
  - Bausch Site 106, Largo, Florida
  - Bausch Site 117, Tampa, Florida
  - Bausch Site 108, Lake Villa, Illinois
  - Bausch Site 112, Indianapolis, Indiana
  - Bausch Site 119, Edgewood, Kentucky
  - Bausch Site 126, Winchester, Massachusetts
  - Bausch Site 113, Kansas City, Missouri
  - Bausch Site 111, St Louis, Missouri
  - Bausch Site 128, Slingerlands, New York
  - Bausch Site 114, Raleigh, North Carolina
  - Bausch Site 122, Cranberry Township, Pennsylvania
  - Bausch Site 107, Memphis, Tennessee
  - Bausch Site 109, Nashville, Tennessee
  - Bausch Site 120, El Paso, Texas
  - Bausch Site 104, Lakeway, Texas
  - Bausch Site 105, Round Rock, Texas
  - Bausch Site 118, San Antonio, Texas

REFERENCES:
- [Derived] Fahmy AM, Harthan JS, Evans DG, Greiner JV, Tauber J, Sheppard JD, Krosser S, Vittitow JL. Perfluorohexyloctane ophthalmic solution for dry eye disease: pooled analysis of two phase 3 clinical trials. Front Ophthalmol (Lausanne). 2024 Nov 5;4:1452422. doi: 10.3389/fopht.2024.1452422. eCollection 2024. PMID 39564145
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NOV03 4 Times Daily (QID) | Placebo 4 Times Daily (QID)
Started | 303 | 294
Completed | 289 | 279
Not Completed | 14 | 15
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lost to Follow-up | 2 | 5
Not completed — Discontinued | 4 | 2
Not completed — Adverse Event | 1 | 3
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NOV03 4 Times Daily (QID) | Placebo 4 Times Daily (QID) | Total
Number analyzed (Participants) | 303 | 294 | 597
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (14.23) | 61.6 (13.57) | 60.9 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219 | 214 | 433
  Male | 84 | 80 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 51 | 94
  Not Hispanic or Latino | 260 | 243 | 503
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFB) in Total Corneal Fluorescein Staining (tCFS) at Day 57
Description: Corneal Fluorescein Staining (tCFS) is graded based on the NEI scale. The NEI scale divides the cornea in 5 subregions: central, inferior, superior, nasal, temporal. The score for each region ranges from 0-3; 0 corresponds to no staining, 3 corresponds to maximum staining. The total score is the sum of the 5 subregions ranging from 0-15.
Time Frame: Assessed from Baseline to Day 57
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | NOV03 4 Times Daily (QID) | Placebo 4 Times Daily (QID)
Number analyzed (Participants) | 289 | 279
Number analyzed (Eyes) | 289 | 279
units on a scale | -2.0 (2.6) | -1.0 (2.7)

2. Primary Outcome: Change From Baseline of Dryness Score at Day 57
Description: Dryness Score is rated on a visual analogue scale (VAS) ranging from 0-100; 0 corresponds to no discomfort and 100 to maximum discomfort).
Time Frame: Assessed from Baseline to Day 57
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | NOV03 4 Times Daily (QID) | Placebo 4 Times Daily (QID)
Number analyzed (Participants) | 289 | 279
Number analyzed (Eyes) | 289 | 279
units on a scale | -27.4 (27.9) | -19.7 (26.7)

ADVERSE EVENTS:
Time Frame: Assessed throughout the study, approximately 8 weeks.
Description: Ocular Treatment-emergent Adverse Events
Arm/Group | NOV03 4 Times Daily (QID) | Placebo 4 Times Daily (QID)
All-Cause Mortality (participants affected / at risk) | 0/303 | 0/294
Serious Adverse Events (participants affected / at risk) | 0/303 | 0/294
Other Adverse Events (participants affected / at risk) | 16/303 | 11/294
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NOV03 4 Times Daily (QID) (N=303) | Placebo 4 Times Daily (QID) (N=294)
Vision blurred (Eye disorders) | 9 | 1
Instillation site pain (Eye disorders) | 3 | 3
Conjunctival haemorrhage (Eye disorders) | 1 | 4
Eye discharge (Eye disorders) | 3 | 0
Punctate keratitis (Eye disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT04139798/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT04139798/SAP_001.pdf